CLINICAL TRIAL: NCT07051213
Title: The Belgian Genome Resource to Resolve Rare Diseases
Acronym: BeSolveRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Erasme University Hospital (Other); University Ghent (Other); Universiteit Antwerpen (Other); Université de Liège (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Institut de Pathologie et de Génétique Charleroi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S64603
Record Dates: First submitted 2025-06-16; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Intellectual Developmental Disorder; Malformations; Dysmorphia; Developmental Delay (Disorder)
Keywords: Whole Genome Sequencing; Whole Exome Sequencing; Rare Disease
MeSH Terms: conditions — Intellectual Disability; Congenital Abnormalities; Developmental Disabilities; Rare Diseases | interventions — Exome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care including Whole Exome Sequencing (Active Comparator): Standard of care consisting of a combination of a chromosomal microarray or shallow whole genome sequencing (standard of care copy number variant analysis in the concerned genetic center) with whole exome sequencing.
  Interventions: Diagnostic Test: Whole exome sequencing
- Whole Genome Sequencing (Experimental): Whole genome sequencing (primary analysis using a similar pipeline as the one used for whole exome sequencing - re-analysis using Emedgene to detect potential repeat expansions, structural and/or intronic variants)
  Interventions: Diagnostic Test: Whole genome Sequencing

INTERVENTIONS:
Diagnostic Test: Whole exome sequencing — Whole exome sequencing using Illumina short read sequencing
  Arms: Standard of Care including Whole Exome Sequencing
Diagnostic Test: Whole genome Sequencing — Whole genome sequencing using Illumina short read sequencing
  Arms: Whole Genome Sequencing

SUMMARY:
Whole-exome (WES) or whole-genome sequencing (WGS) are recommended as first- or second-tier molecular tests for patients with developmental disorders (DD), but the clinical utility of WGS continues to be debated. This prospective randomized trial involving all Belgian Human Genetics centers compares the standard of care (SoC) - combining WES and microarray or shallow WGS - with WGS for 567 individuals with unexplained DD. The aim of the project is to pave the way towards diagnostic implementation of WGS for rare DD in Belgium. To reach this aim, (1) technical validation is performed at different genetic centres in Belgium, (2) clinical utility of WGS is explored and (3) the health economic impact is mapped.

ELIGIBILITY:
Inclusion Criteria:

* Intellectual disability/Developmental delay (moderate to profound)
* Intellectual disability/Developmental delay (mild to moderate) AND family recurrence AND normal parents
* Intellectual disability/Developmental delay (mild to moderate) AND dysmorphism (≥3 well documented minor signs)
* One major malformation AND dysmorphism (≥3 well documented minor signs)
* Multiple major malformations in 2 or more different organ systems.

Exclusion Criteria:

* Suspicion of an acquired cause, e.g. congenital infection and prenatal toxic exposure
* Prior next-generation sequencing of a gene panel targeting multiple conditions or prior exome analyses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Whole genome sequencing (WGS) performance compared to Whole exome sequencing (WES) performance | From enrollment to reporting the results of the analysis : target turn around time of 6 months
  The primary outcome measure is to determine whether whole genome sequencing is able to improve the diagnostic yield of next-generation sequencing for developmental disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The raw sequencing data generated during this study will be shared on the European Genome-phenome Archive (EGA).